CLINICAL TRIAL: NCT06107842
Title: Relationship of Exercise Frequency, Intensity, and Fitness to Improved Cognition and Biomarkers in Gerofit Participants
Brief Title: Gerofit and Cognition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E4521-R
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Aging; Cognitive Impairment; Physical Activity
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: Gerofit intervention vs Health Education Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gerofit exercise (Active Comparator): Participants enrolled in the Gerofit program
  Interventions: Behavioral: Gerofit exercise
- Health education (Placebo Comparator): Participants enrolled in monthly in-person health education sessions which do not include a physical activity/exercise promotion session
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Gerofit exercise — Individualized exercise prescription as well as a group exercise class based on physical function assessments offered 3x/week
  Arms: Gerofit exercise
Behavioral: Health education — Scheduled monthly in-person health education discussion sessions covering 12 different health topics not including a physical activity/exercise promotion session
  Arms: Health education

SUMMARY:
Over 50% of the Veterans enrolled for VA health care are over the age of 65. Dementia prevalence increases with age, and with the increase in the population of people ages 65 and older, the total number of people with dementia is also increasing. Older Veterans often have comorbid PTSD, major depression and traumatic brain injury so that they are at 2 to 5 times the risk for cognitive impairment and dementia compared to the general population. There is evidence that exercise interventions in sedentary older adults could improve both physical and cognitive function. However, there have been very few studies on the effects of exercise on cognition in older Veterans and do not reflect the broader ethnic and health-status diversity of Veterans. Thus, improved knowledge of the role of exercise on cognition as well as the predictive power of biomarkers could have a major beneficial impact on Veterans' functional independence and quality of life. The investigators hypothesize that participation in the VA Gerofit exercise program will improve cognitive function in older Veterans and that blood and muscle biomarkers will predict these improvements.

ELIGIBILITY:
Inclusion Criteria:

* All Veterans eligible for VA Gerofit program 65 years and older
* Clearance by PCP to participate in Gerofit exercise program

Exclusion Criteria:

* Inability to perform ADLs
* Significant cognitive impairment
* Inability to function independently without assistance
* Unstable angina; proliferative diabetic retinopathy
* Oxygen dependent
* Unwillingly to commute and/or not able to provide own transportation to Gerofit
* Incontinence
* Open wounds
* Volatile behavioral issue or unable to work successfully in a group environment/setting
* Active substance abuse
* Homelessness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Memory composite score | Change from baseline at 3 months
  HVLT-R, verbal memory and BVMT-R, visual memory
Executive Function composite score | Change from baseline at 3 months
  Stroop C, Trails B, Digit span backwards and sequencing from WAIS-IV, verbal fluency, FAS and animals
Total BDNF | Change from baseline at 3 months
  Total brain derived neurotrophic factor (BDNF) concentrations in serum
Mature BDNF | Change from baseline at 3 months
  Mature brain derived neurotrophic factor (BDNF) concentrations in serum
Memory composite score | Change from baseline at 12 months
  HVLT-R, verbal memory and BVMT-R, visual memory
Executive Function composite score | Change from baseline at 12 months
  Stroop C, Trails B, Digit span backwards and sequencing from WAIS-IV, verbal fluency, FAS and animals
Total BDNF | Change from baseline at 12 months
  Total brain derived neurotrophic factor (BDNF) concentrations in serum
Mature BDNF | Change from baseline at 12 months
  Mature brain derived neurotrophic factor (BDNF) concentrations in serum

CONTACTS AND LOCATIONS:
Overall Officials: Cathy C Lee, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Jonathan M Wanagat, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Stacy Wilkins, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No